CLINICAL TRIAL: NCT00005415
Title: Physical Activity Effects on Health Care Utilization
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4333; R03HL047519 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2000-06

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

SUMMARY:
To determine the magnitude of the relationship between physical activity level and subsequent health care utilization over a seven to ten week period in a general population.

DETAILED DESCRIPTION:
BACKGROUND:

In recent years, the benefits of a physically active lifestyle have been well established with respect to chronic health problems such as coronary heart disease, hypertension, obesity and osteoporosis. However, the extent to which physical activity influences health care utilization is less clear. If physical activity levels are inversely associated with utilization patterns, then policies encouraging exercise may produce short-term reduction in health care costs.

DESIGN NARRATIVE:

A multivariate regression analysis was conducted for a representative sample of more than 600 adults who participated in a longitudinal field trial of health risk appraisal instruments. Using the Harvard Alumni Activity Survey as the physical activity measure, the analysis controlled for a variety of predisposing, enabling, and need characteristics that also influenced utilization behavior.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1992-09; Study Completion 1993-09 (Actual)